CLINICAL TRIAL: NCT02319915
Title: Evaluation of the Pharmacokinetic Profile of Tranexamic Acid, After Injection in a Knee Neo-articulation.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Philippe VAN DER LINDEN, Pr, MD, Head of clinic, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHUB-PTGexacyl-001
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Knee Prosthesis
Keywords: tranexamic acid; knee prosthesis; pharmacokinetic profile
MeSH Terms: interventions — Tranexamic Acid; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic acid (Experimental): Study of the pharmacokinetic profile of the plasmatic resorption of tranexamic acid after an intra-articular injection.
  Interventions: Drug: Tranexamic Acid
- Tranexamic acid + adrenalin (Active Comparator): Study of the pharmacokinetic profile of the plasmatic resorption of tranexamic acid after an intra-articular injection of tranexamic acid with adrenalin 1/200 000.
  Interventions: Drug: Tranexamic Acid; Drug: Adrenalin

INTERVENTIONS:
Drug: Tranexamic Acid
Drug: Adrenalin
  Arms: Tranexamic acid + adrenalin

SUMMARY:
Evaluate the pharmacokinetic profile of tranexamic acid injected intra-articularly with or without adrenaline, in a population of patients undergoing knee replacement.

DETAILED DESCRIPTION:
Orthopedic population, especially during a knee surgery, is at risk of significant bleeding and blood transfusion in the perioperative period. Tissue damage is associated with the activation of a cascade of mechanisms, in which the activation of the fibrinolyse plays an important role. This is why anti-fibrinolytic agents are regularly used in this context to reduce the perioperative bleeding and the use of blood transfusions.

In the majority of cases, tranexamic acid, an analogue agent of lysine, is administered by an intravenous injection and more recently, by an intra-articular injection.

Several questions however remain unanswered.

* what is the clearance of this substance ?
* does an intra-articular resorbtion exist, resulting in a plasmatic rate of the substance ? If yes, what is the plasmatic rate ?
* Is the intra-articular effect of tranexamic acid predominant compared to its systemic effect ?
* Does the addition of adrenalin increase the effect of the tranexamic acid by acting on its absorption ?

The efficacy, safety and better administration route of the tranexamic acid remain unknown when injected intra-articularly. The goal of this study is to realize the first pharmacokinetic study after an intra-articular injection of tranexamic acid, alone of along with adrenalin, in a knee neo-articulation.

ELIGIBILITY:
Inclusion Criteria:

* programmed PTG, right or left
* surgery planned within the CHU Brugmann Hospital (Dr Reynders)
* ASA I to ASA III
* Signed informed consent within the patient file

Exclusion Criteria:

* re-do surgery
* urgent or multiple surgery
* ASA IV or higher
* Patients with a BMI superior or equal to 40
* Patient is a Jehovah Witness
* Allergy or contra-indication to tranexamic acid
* Coagulation troubles, defined as: Platelet count < 80 000/mm3 and/or PTT <70% and/or aPTT >45s and/or Fibrinogen <100mg/dL
* Preoperatory renal insufficiency defined as Creatinin > 3mg/dL and/or Dialysis patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-02-18 (Actual); Primary Completion 2017-03-14 (Actual); Study Completion 2017-03-14 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic profile of tranexamic acid | 24h
  Blood sampling will be performed to establish the pharmacokinetic profile of tranexamic acid. T0 will be defined as the injection time of tranexamic acid. The first blood sampling (T1) will be made 5 minutes after, with the garrot still in place. The garrot will then be loosened and the following blood samplings will take place at 1 minute, 5 minute, 15 minutes, 30 minutes, 1h, 2h, 4h, 8h, 12h and 24h after garrot loosening. 1ml of blood will be taken at each blood sampling. The blood will be placed in a tube suited for chemistry analysis (green tube with gel) and sent directly to the laboratory for analysis.

SECONDARY OUTCOMES:
Knee diameter | 12h
  This will be part of the semi-quantitative evaluation of the knee bleeding. The diameter of both knees (the one undergoing surgery and the untouched one) will be measured before and after surgery.
Net weight of the compresses | 12h
  This will be part of the semi-quantitative evaluation of the knee bleeding. The net weight of the blood soaked compresses will be measured.
Size of the blood stain on the band aid | 12h
  This will be part of the semi-quantitative evaluation of the knee bleeding. The size of the blood stain, defined as the percentage of the circumference of the band aid that is blood stained, will be measured.
Blood loss | 72h
  The blood loss will be deduced from the estimated circulating volume and the patient hematocrit level before and 72h after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Van der Linden, MD, Pr, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Gandhi R, Evans HM, Mahomed SR, Mahomed NN. Tranexamic acid and the reduction of blood loss in total knee and hip arthroplasty: a meta-analysis. BMC Res Notes. 2013 May 7;6:184. doi: 10.1186/1756-0500-6-184. PMID 23651507
- [Background] Chareancholvanich K, Siriwattanasakul P, Narkbunnam R, Pornrattanamaneewong C. Temporary clamping of drain combined with tranexamic acid reduce blood loss after total knee arthroplasty: a prospective randomized controlled trial. BMC Musculoskelet Disord. 2012 Jul 20;13:124. doi: 10.1186/1471-2474-13-124. PMID 22817651
- [Background] Ortega-Andreu M, Perez-Chrzanowska H, Figueredo R, Gomez-Barrena E. Blood loss control with two doses of tranexamic Acid in a multimodal protocol for total knee arthroplasty. Open Orthop J. 2011 Mar 16;5:44-8. doi: 10.2174/1874325001105010044. PMID 21552468
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Mutsuzaki H, Ikeda K. Intra-articular injection of tranexamic acid via a drain plus drain-clamping to reduce blood loss in cementless total knee arthroplasty. J Orthop Surg Res. 2012 Sep 29;7:32. doi: 10.1186/1749-799X-7-32. PMID 23020868
- [Background] Sa-Ngasoongsong P, Channoom T, Kawinwonggowit V, Woratanarat P, Chanplakorn P, Wibulpolprasert B, Wongsak S, Udomsubpayakul U, Wechmongkolgorn S, Lekpittaya N. Postoperative blood loss reduction in computer-assisted surgery total knee replacement by low dose intra-articular tranexamic acid injection together with 2-hour clamp drain: a prospective triple-blinded randomized controlled trial. Orthop Rev (Pavia). 2011;3(2):e12. doi: 10.4081/or.2011.e12. Epub 2011 Jun 29. PMID 22053253
- [Background] Ishida K, Tsumura N, Kitagawa A, Hamamura S, Fukuda K, Dogaki Y, Kubo S, Matsumoto T, Matsushita T, Chin T, Iguchi T, Kurosaka M, Kuroda R. Intra-articular injection of tranexamic acid reduces not only blood loss but also knee joint swelling after total knee arthroplasty. Int Orthop. 2011 Nov;35(11):1639-45. doi: 10.1007/s00264-010-1205-3. Epub 2011 Jan 21. PMID 21253725
- [Background] Samama CM, Langeron O, Rosencher N, Capdevila X, Rouche P, Pegoix M, Berniere J, Coriat P. Aprotinin versus placebo in major orthopedic surgery: a randomized, double-blinded, dose-ranging study. Anesth Analg. 2002 Aug;95(2):287-93, table of contents. doi: 10.1097/00000539-200208000-00005. PMID 12145035